CLINICAL TRIAL: NCT03426982
Title: A Randomized Study Aimed at Comparing Activated Partial Thromboplastin Time and Anti-Xa Activity and in Patients Requiring Unfractionated Heparin Infusion
Brief Title: Comparision Between Activated Partial Thromboplastin Time Versus Anti-Xa Activity in Heparin Monitoring
Acronym: CATCH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan Asia Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-P-002
Record Dates: First submitted 2018-02-01; First posted 2018-02-09 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Myocardial Infarction; Venous Thromboembolism; Stroke; Bleeding
MeSH Terms: conditions — Myocardial Infarction; Venous Thromboembolism; Stroke; Hemorrhage | interventions — Heparin

STUDY DESIGN:
Intervention Model Description: After randomization, the patients must be monitored using either anti-Xa activity or aPTT.
  Only that specific test should be prescribed by the ward, and only that the corresponding test result be given by the laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-Xa group (Experimental): - Heparin was monitored by Anti-Xa activity, and clinicians adjusted dose of heparin to maintain it within the therapeutic range between 0.30 and 0.70 IU/mL
  Interventions: Drug: Unfractionated heparin
- APTT group (Experimental): - Heparin was monitored by APTT, and clinicians adjusted dose of heparin to maintain it within the therapeutic range between 1.5 and 2.5 time the basiline.
  Interventions: Drug: Unfractionated heparin

INTERVENTIONS:
Drug: Unfractionated heparin — Infusion dose of unfractionated heparin was adjusted by APTT
  Arms: APTT group
Drug: Unfractionated heparin — Infusion dose of unfractionated heparin was adjusted by anti-Xa
  Arms: Anti-Xa group

SUMMARY:
Background:

Unfractionated heparin (UFH) is a sulfated polysaccharide extracted from porcine intestinal mucosa that enhances the inhibitory activity of the natural anticoagulant antithrombin towards most activated clotting factors (F), particularly FXa and FIIa (thrombin) . Despite the growing interest for low molecular weight derivatives (LMWH), UFH is still widely used for different indications including the treatment of acute thrombosis including venous thromboembolism, coronary syndromes (ACS), and other thrombotic diseases. UFH is administered by parenteral route either intravenous (IV) or sub-cutaneous (SC).Actually, there is evidence that the risk of recurrence of thrombosis is increased when heparin levels fells below the lower limit of the therapeutic range, while the hemorrhagic risk increases with heparin levels above the upper limit of the therapeutic range. Moreover, the anticoagulant response to UFH is highly variable for one individual to another. As the clinical efficacy of heparin is dependent on maintaining an anticoagulant effect above a minimum level, careful laboratory monitoring of UFH treatment is mandatory. For that purpose, two options are offered to the clinicians: i) to evaluate either the prolongation of a global clotting assay, the activated partial thromboplastin time (aPTT) and ii) to measure the heparin-enhanced inhibitory activity of AT toward purified activated factors such as FIIa and FXa using chromogenic substrate-based assays. UFH therapy is still widely monitored by the aPTT, a global clotting assay, that reflects the ability of heparin to enhance the inhibitory activity of AT against FIIa, FXa, and other activated factors. The therapeutic range of aPTT prolongation is highly dependent on the reagent and analyzer used. As the consequence, it must be defined by each laboratory in its own technical conditions (for each reagent batch) to correlate with heparin levels between 0.20 and 0.40 U/mL (protamine sulfate titration), corresponding to anti-FXa activity between 0.30 and 0.70 IU/mL. In that connection, the prolongation of aPTT corresponding to antiFXa activity between 0.30 - 0.70 IU/mL is highly variable depending of the reagents e.g.between 1.6 - 2.7 x control for weakly sensitive reagents and between 3.7 - 6.2 x control for highly sensitive reagents. The use of aPTT has advantages as it is easy-to-perform, quick, inexpensive but faces numerous challenges due to the significant influence of the technical conditions (reagent/instrument) on the test result, to lot-lot variation in reagent sensitivity, to the need of studies to evaluate the therapeutic range, to limited therapeutic range, and also to non-specific prolongation in the case of lupus anticoagulant, factors deficiency, inhibitors or shortening in the case of high factor levels, particularly FVIII.In contrast, the use of chromogenic anti-Xa assays has many advantages particularly a published therapeutic range for UFH i.e. between 0.30 and 0.70 IU/mL, a specificity to its interaction with AT (no Heparin Cofactor II interference by using bovine FIIa or short incubation time) and faces few challenges such as limited availability in some area and a cost that is slightly higher than that of aPTT. In addition, anti-Xa assays allow accurate measurement of all heparin(s) derivatives and particularly LMWHs and fondaparinux.

Since the first reports in the mid-eighties, some small sized studies have compared the two monitoring strategies mainly retrospectively designed (7-11). Even though, one single prospective randomized management study evaluated the comparison between the two monitoring strategies with clinical end-points i.e. recurrence of thrombosis and bleeding complication in a cohort of 131 patients with VTE . All concluded to a trend toward higher, or at least similar, safety/efficacy/efficiency when patients were monitored using antiXa activity vs. aPTT. Even though differences were not significant due to the lack of power of these studies.

DETAILED DESCRIPTION:
Aim of the study Based on available data, a randomized trial aimed at comparing the efficacy and safety of monitoring UFH treatments using aPTT and anti-FXa activity in patients treated with fulldoses of UFH could validly be carried out.

Study design

* Primary objectives: safety and efficacy
* Secondary objectives: efficiency and cost effectiveness
* Primary evaluation criteria: bleeding complications (n, %) and thrombotic complications
* Secondary evaluation criteria: percentage of test results within the therapeutic range,number of tests perfomed per day, number of daily dose adjustments, total dosage of heparin given to the patients, mean time to achieve therapeutic anticoagulation, transfusion rates, health economics analysis (total treatment cost)
* Calculation of number of patients to be evaluated:

According to the only randomized study published to date (A), the bleeding rate was 1.5% (n=1/65) in the group of patients monitored using Anti-FXa activity vs. 6.1% (n=4/66) in theaPTT group. The difference was not significant (p=0.36) due to the lack of power of the study (n=131 patients). Taking into account these bleeding risks and 0.05 as the alpha risk and 0.20 (0.05) as the beta risk, the number of patients to be included would be 323 (506) in each treatment arm.

Description of the two monitoring strategies

Patients should be randomized to be monitored using either:

* Anti-Xa activity (heparin levels) with the therapeutic range between 0.30 and 0.70IU/mL (corresponding to 0.2 to 0.4 protamine sulfate titration assay) (3).
* aPTT wIth the usual therapeutic range of 1.5 to 2.5 fold the control time, which was the usually used therapeutic range in the institution.

Example of nomogram for heparin dose-adjustment when monitored using aPTT or anti-Xa activity (12)Practical considerations

* Mechanism of randomization: electronic
* After randomization, the patients must be monitored using either anti-Xa activity or aPTT.

Only that specific test should be prescribed by the ward, and only that the corresponding test result be given by the laboratory.

* Ideally, fresh patients samples should be evaluated for both Anti-Xa activity and aPTT, data being recorded, but only the prescribed test should be given to the ward. In addition, it would be necessary to store aliquots (0.5-1.0 mL each) of plasmas samples frozen at -70°C for control purpose.
* Patients must be follow-up at 3-months
* Data to be collected:

Patients demographical data (sex, age), indication of UFH therapy (VTE, ACS, other…),comorbidity (cancer, pregnancy, postoperative period, other…), concomitant therapy (medication such as oral contraceptive…) , previous history of thrombosis (DVT, ACS,stroke, other…) Duration (in hours) and total dosage (IU) of heparin therapy before randomization (if any) Route of administration (IV, SC), daily heparin dosage (IU), duration of treatment, time to achieve therapeutic range, number of dosage change per day, laboratory test results (anti-Xa activity or aPTT) Outcome: death (any cause (to be recorded), description of any bleeding complication (when, localization, classification as major or minor…) or recurrence of thrombosis (when,localization…) while on UFH therapy and within the 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* acute venous thromboembolism,
* acute coronary syndrome
* receiving UFH therapy.

Exclusion Criteria:

* non-willing to participate in the study,
* thrombolytic therapy,
* previous treatment with heparin (UFH) of more than one day before randomization,
* history of heparin-induced thrombocytopenia.
* other conditions considering by study clinians that are not suitable for the trail.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Bleeding | 30 days
  Any bleeding events including major bleeding and minor bleeding
Ischemic vascular events | 30 days
  Repeat MI, recurrence of thrombosis

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Asia Heart Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided